CLINICAL TRIAL: NCT01713933
Title: Evaluation of the Ulthera® System for Obtaining Lift and Tightening of the Brachia
Brief Title: Evaluation of the Ulthera® System for Treatment of the Brachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-114
Record Dates: First submitted 2012-10-15; First posted 2012-10-25 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Brachial Ptosis
Keywords: Ulthera® System; Ultherapy™ treatment; Ulthera, Inc.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy™ treatment (Experimental): Each enrolled subject will receive a bilateral Ultherapy™ treatment of the upper arms
  Interventions: Device: Ulthera® System

INTERVENTIONS:
Device: Ulthera® System — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy™ treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening

SUMMARY:
This study is an evaluation of the Ulthera® System used to treat the upper arms for improvement of brachial ptosis. All enrolled subjects will receive one bilateral upper arm treatment. Follow-up visits will occur at 60, 90 and 180 days post-treatment.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, clinical trial treating up to 35 subjects. Study photographs of the upper arms will be taken prior to treatment, immediately post-treatment, and at each follow-up visit. Brachial volume and dermal thickness measurements will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 19 - 55 years.
* Subject in good health.
* Subjects who desire lift and tightening of the brachia and improvement in skin laxity.
* Mild to moderate laxity of the upper arm.
* Mild to moderate subcutaneous fat of the upper arm.
* Mild crepiness of the skin of the upper arm.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the upper arm.
* Excessive skin laxity in the upper arm.
* Significant scarring in areas to be treated.
* Significant open wounds or lesions in the treatment areas. 7. Severe or cystic acne in the treatment areas.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Sasaki, MD FACS, Principal Investigator — Sasaki Advanced Aesthetic Medical Center
Locations (1):
- Sasaki Advanced Aesthetic Medical Center, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened 6/29/2011 and the last subject was treated 11/28/2011. Subjects were recruited from the site's patient database.
Groups:
- Ultherapy® Treatment: Each enrolled subject will receive a bilateral Ultherapy® treatment of the upper arms
Period: Overall Study
Arm/Group | Ultherapy® Treatment
Started | 37
Completed | 31
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Excluded from analysis as a BMI outlier | 1

BASELINE CHARACTERISTICS:
Population: Three subjects excluded due to subject withdrawal. One subject excluded from results analyses as an outlier, with a high Body Mass Index (BMI) and substantial weight gain during the study period.
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 40 [25 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 33
Fitzpatrick Skin Type [Number; unit: Participants] — Skin Type I = White;very fair,red or blonde hair blue eyes;freckles;Always burns, never tans Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes;Usually burns, tans with difficulty Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily Skin Type VI = Black; Never burns, tans very easily
  Participants
    Type I | 0
    Type II | 0
    Type III | 15
    Type IV | 16
    Type V | 2
    Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Obtaining Lift and Tightening of Brachial Skin Laxity
Description: Improvement in overall lifting and tightening of brachial skin laxity as determined by masked, qualitative assessment of photographs at 90 days post-treatment compared to baseline.
Time Frame: Baseline to 90 days post-treatment
Population: Twenty-seven (27) subjects returned for the 90 day post-treatment visit. Five (5) 90 day visits were missed, including the one subject excluded from analyses as an outlier due to high Body Mass Index (BMI) and substantial weight gain during the study period. Two (2) subjects were lost-to-follow-up.
Measure: Number; unit: percentage of participants improved
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 27
percentage of participants improved | 48

2. Secondary Outcome: Quantitative Improvement in Skin Laxity
Description: Assess change in brachial volume based on brachial tissue measurements.
Time Frame: Baseline to 90 days post-treatment
Population: Twenty-seven (27) subjects returned for the 90 day post-treatment visit. Five (5) 90 day visits were missed, including one subject excluded from analyses as an outlier due to high BMI and substantial weight gain during the study period. Two (2) subjects were lost-to-follow-up.
Measure: Number; unit: percentage of participants improved
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 27
percentage of participants improved
  Improvement Left Arm | 54
  Improvement Right Arm | 62
  Improvement of both Left & Right Arms | 35

3. Secondary Outcome: Change in Dermal Thickness
Description: Based on ultrasonic skin analysis, the change in dermal thickness from baseline to 90 days post-treatment was calculated.
Time Frame: Baseline to 90 days post-treatment
Population: as for outcome 2
Measure: Mean (Full Range); unit: Millimeters
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 27
Millimeters
  Difference in Mean Thickness from Baseline - R Arm | 0.072 [-0.015 to 0.224]
  Difference in Mean Thickness from Baseline - L Arm | 0.082 [-0.170 to 0.296]

4. Secondary Outcome: Change in Dermal Thickness
Description: Based on ultrasonic skin analysis, the change in dermal thickness from baseline to 180 days post-treatment was calculated.
Time Frame: Baseline to180 days post-treatment
Population: Thirty-one (31) subjects returned for the 180 day post-treatment visit. Two subjects were lost-to-follow-up. One subject was excluded from analyses as an outlier due to high BMI and substantial weight gain during the study period.
Measure: Mean (Full Range); unit: Millimeters
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 31
Millimeters
  Difference in Mean Thickness from Baseline - R Arm | 0.099 [0.002 to 0.330]
  Difference in Mean Thickness from Baseline - L Arm | 0.085 [0.034 to 0.459]

5. Secondary Outcome: Overall Aesthetic Improvement
Description: Based on Global Aesthetic Improvement Scale (GAIS) Scores; PGAIS completed by a physician assessor, SGAIS completed by the study subject. . The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse
Time Frame: Baseline to 60 days post-treatment
Population: Thirty-one (31) subjects returned for the 60 day post-treatment visit. Two subjects were lost-to-follow-up. One subject was excluded from analyses as an outlier due to high BMI and substantial weight gain during the study period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 31
Percentage of Participants
  Subject GAIS Very Much Improved | 0
  Subject GAIS Much Improved | 0
  Subject GAIS Improved | 51.6
  Subject GAIS No Change | 48.4
  Subject GAIS Worse | 0
  Physician GAIS Very Much Improved | 0
  Physician GAIS Much Improved | 0
  Physician GAIS Improved | 67.7
  Physician GAIS No Change | 32.2
  Physician GAIS Worse | 0

6. Secondary Outcome: Overall Aesthetic Improvement
Description: as for outcome 5
Time Frame: Baseline to 90 days post-treatment
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 27
Percentage of Participants
  Subject GAIS Very Much Improved | 0
  Subject GAIS Much Improved | 3.7
  Subject GAIS Improved | 59.3
  Subject GAIS No Change | 37.0
  Subject GAIS Worse | 0
  Physician GAIS Very Much Improved | 0
  Physician GAIS Much Improved | 0
  Physician GAIS Improved | 66.6
  Physician GAIS No Change | 33.3
  Physician GAIS Worse | 0

7. Secondary Outcome: Overall Aesthetic Improvement
Description: as for outcome 5
Time Frame: Baseline to180 days post-treatment
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 31
Percentage of Participants
  Subject GAIS Very Much Improved | 6.5
  Subject GAIS Much Improved | 16.1
  Subject GAIS Improved | 48.4
  Subject GAIS No Change | 29
  Subject GAIS Worse | 0
  Physician GAIS Very Much Improved | 0
  Physician GAIS Much Improved | 19.4
  Physician GAIS Improved | 61.3
  Physician GAIS No Change | 19.4
  Physician GAIS Worse | 0

8. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was determined by scores on a patient satisfaction questionnaire (PSQ) completed at 90 days post-treatment. Subjects indicated how satisfied they were with study treatment, i.e., Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Pre-treatment and Day 90 post-treatment photographs were available for viewing during the assessment.
Time Frame: Baseline to 90 days post-treatment
Population: wenty-seven (27) subjects returned for the 90 day post-treatment visit. Five (5) 90 day visits were missed, including one subject excluded from analyses as an outlier due to high BMI and substantial weight gain during the study period. Two (2) subjects were lost-to-follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 27
Percentage of Participants
  Very Satisfied | 14.8
  Satisfied | 59.2
  Dissatisfied | 22.2
  Very Dissatisfied | 3.7
  Improvement Noticed | 55.5

9. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was determined by scores on a patient satisfaction questionnaire (PSQ) completed at 180 days post-treatment. Subjects indicated how satisfied they were with study treatment, i.e., Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Pre-treatment and Day 90 post-treatment photographs were available for viewing during the assessment.
Time Frame: Baseline to 180 days post-treatment
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Ultherapy® Treatment
Number analyzed (Participants) | 31
Percentage of Participants
  Very Satisfied | 12.9
  Satisfied | 64.5
  Dissatisfied | 22.5
  Very Dissatisfied | 0
  Improvement Noticed | 70.9

ADVERSE EVENTS:
Arm/Group | Ultherapy® Treatment
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

LIMITATIONS AND CAVEATS:
- Poor subject selection (high BMI with large volume arms enrolled rather than subjects with laxity and wrinkled skin)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less